CLINICAL TRIAL: NCT07029984
Title: Baylor Continence Scale in Children With Anorectal Malformations: A Turkish Validity and Reliability Study
Brief Title: Baylor Continence Scale Validity in Anorectal Malformation
Status: Recruiting | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, AYŞE KAYALI VATANSEVER, Assistant Professor, PhD, Izmir Bakircay University
Other Study IDs: 2015
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Validity and Reliability Study in Children With Anorectal Malformations
Keywords: Anorectal Malformation; Baylor Continence Scale; Validity and Reliability
MeSH Terms: conditions — Anorectal Malformations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Anorectal Malformations: Having undergone surgery due to anorectal malformations, Being between 6 and 18 years of age, The child and caregiver knowing Turkish
  Interventions: Other: Baylor Continence Scale

INTERVENTIONS:
Other: Baylor Continence Scale — This study may be one of the first to test the Turkish adaptation and validity of the scale in Turkish children with anorectal malformations.

SUMMARY:
The aim of this study is to evaluate the validity and reliability of the Baylor Continence Scale in Turkish-speaking children diagnosed with anorectal malformations. The scale is used to assess continence levels, helping healthcare providers make informed decisions regarding treatment and follow-up. The study includes a sample of children with confirmed anorectal malformations, and data collection consists of language adaptation, statistical validation, and reliability testing. Results will contribute to the standardization of continence assessment in Turkish clinical settings, ensuring accurate evaluations for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone surgery due to anorectal malformation
* Being between 6 and 18 years old
* The child and caregiver are required to know Turkish

Exclusion Criteria:

* The child and caregiver having comprehension, hearing, or vision problems

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Inclusion criteria for the study include children who have undergone surgery due to anorectal malformation, are between 6 and 18 years old. Exclusion criteria consist of cases where the child and caregiver have comprehension, hearing, or vision problems that could affect communication or participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Validity and Reliability Analyses | Average 6 to 12 month
  In this study, validity and reliability analyses will be conducted as part of the Turkish adaptation of the Baylor Continence Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Department of Pediatric Surgery and Bakırçay University Physical Therapy and Rehabilitation Application and Research Center, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No